CLINICAL TRIAL: NCT05098145
Title: A Single-arm, Multi-center, Open-label Proof of Concept Safety and Efficacy Study of FCR001 Cell-based Therapy in Adults With Rapidly Progressive Diffuse Cutaneous Systemic Sclerosis at Risk for Organ Failure
Brief Title: A Safety and Efficacy Study of FCR001 in Adults With Rapidly Progressive Diffuse Cutaneous Systemic Sclerosis
Acronym: FREEDOM-3
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: all clinical development programs terminated by sponsor
Sponsor: Talaris Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FCR001C2201 (FREEDOM-3)
Record Dates: First submitted 2021-10-20; First posted 2021-10-28 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Diffuse Cutaneous Systemic Sclerosis
Keywords: Stem cell therapy; Scleroderma; Severe scleroderma; Allogeneic; Transplant
MeSH Terms: conditions — Scleroderma, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- FCR001 (Experimental): FCR001 is a cryopreserved allogeneic stem cell therapy derived from mobilized peripheral blood cells and delivered as a single infusion with a nonmyeloablative conditioning regimen.
  Interventions: Biological: FCR001

INTERVENTIONS:
Biological: FCR001 — Enriched hematopoietic stem cell infusion

SUMMARY:
This is a multicenter, open-label study to evaluate the safety and tolerability and explore the efficacy of FCR001 cell therapy in adults with rapidly progressive Diffuse Cutaneous Systemic Sclerosis (dcSSc) at risk for organ failure.

DETAILED DESCRIPTION:
The purpose of this multicenter, single-arm study is to evaluate the safety and tolerability and explore the efficacy of FCR001 cell therapy in adults with rapidly progressive dcSSc at risk for organ failure. It consists of 2 years of treatment and 3 years of follow-up, with the primary analysis performed at 24 months.

FCR001 is a cell therapy product that is administered by intravenous (IV) infusion, following nonmyeloablative (NMA) conditioning. It consists of mobilized peripheral blood cells, facilitating cells, and αβ T cells. This therapy is designed to induce donor-specific tolerance by establishing sustained chimerism and to protect against graft versus host disease (GvHD), the major impediment for advancing allogeneic hematopoietic stem cell therapy (HSCT) as a potential therapy in patients.

ELIGIBILITY:
Key Inclusion Criteria (Recipients):

1. Age ≥ 18 and < 70 years
2. Diagnosis of diffuse cutaneous systemic sclerosis
3. Disease duration < 5 years from first non-Raynaud's phenomenon symptom
4. Received at least one immunosuppressant in the past to treat the systemic sclerosis (SSc) or currently on an immunosuppressive therapy
5. Modified Rodnan Skin Score > 15 and < 40
6. Documented evidence of pulmonary or renal involvement by having at least one of the following:

   a) Pulmonary, both required: i. FVC > 45% and < 80% predicted or hemoglobin-adjusted DLco > 45% and < 80% predicted AND ii. Interstitial lung disease evidenced by chest high-resolution computed tomography b) Renal: history of renal crisis that is not active at time of screening. Stable serum creatinine (< 20% increase) must be documented for a minimum of 3 months post-renal crisis at the time of the screening visit.

Key Inclusion Criteria (Donors): Age ≥ 18 and < 60 years

Key Exclusion Criteria (Donor and Recipient):

1. Use of investigational drugs within 30 days (or within 5 drug half-lives) of signing informed consent
2. Pregnant or nursing (lactating) woman
3. Human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV) positive. Those with history of HCV infection which was successfully treated and cured may participate
4. History of malignancy (other than localized squamous or basal cell carcinoma of the skin or in-situ cervical cancer without recurrence) or premalignant syndrome within the past 5 years
5. Known bone marrow aplasia

Key Exclusion Criteria (Recipient):

1. Rheumatic disease, other than systemic sclerosis
2. FVC < 45% of predicted or hemoglobin-adjusted DLco < 45% of predicted
3. Pulmonary arterial hypertension (PAH)
4. An LVEF < 50% by echocardiogram or clinical evidence of significant CHF (New York Heart Association Class III or IV) or symptomatic cardiac disease or uncontrolled clinically significant arrhythmias
5. Estimated GFR < 40 mL/min
6. Previous treatment with cyclophosphamide, as defined by combination of prior oral and intravenous cyclophosphamide > 9 months, independent of dose
7. Corticosteroid therapy at prednisone equivalent doses of greater than 10 mg/day, or more than two pulses for concurrent illnesses within prior 12 months
8. Uncontrolled hypertension
9. Active gastric antral vascular ectasia, also known as "watermelon stomach"
10. Use of scleroderma specific therapies beyond protocol specified washout period, except for PDE-5 inhibitors for Raynaud's phenomenon and digital ulcers
11. Previous history of bone marrow transplant, total lymphoid irradiation, solid organ transplant, autologous or allogeneic hematopoietic progenitor or mesenchymal stem cell transplant
12. Presence of donor-specific antibodies
13. Body mass index < 18 or > 35 kg/m^2

Key Exclusion Criteria (Donor): Biologically unrelated female donor to male recipient

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-11-24 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of recipient adverse events (AEs) | From day before infusion to 60 months
Incidence of recipient serious adverse events (SAEs) | From day before infusion to 60 months
Occurrence of Graft versus Host Disease (GvHD) | From infusion to 60 months
Time to neutrophil recovery | From infusion to 28 days
Time to platelet recovery | From infusion to 28 days

SECONDARY OUTCOMES:
Percent donor whole blood chimerism | From infusion to 60 months
Percentage of donor T-cell chimerism | From infusion to 60 months
Incidence of donor AEs | From donation to 12 months
Incidence of donor SAEs | From donation to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Joel Weinthal, MD, Study Director — Talaris Therapeutics
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No